CLINICAL TRIAL: NCT03362411
Title: Randomized, Open-Label Study to Assess the Relative Bioavailability of a Single 100-mg Dose of BMS-986205 in Healthy Participants When Administered as a Crushed Tablet Orally or Crushed Tablet Suspension Via Nasogastric Tube Compared to an Intact Tablet of Similar Dose
Brief Title: A Study to Assess the Absorption of a Single Dose of BMS-986205 in Healthy Volunteers When Administered as a Crushed Tablet Orally or Crushed Tablet Suspension Via Nasogastric Tube, as Compared to a Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA017-070
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy participants; Healthy subjects
MeSH Terms: interventions — linrodostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986205 intact tablet orally then crushed tablet orally (Experimental): Single, 100 mg dose
  Interventions: Drug: BMS-986205
- BMS-986205 crushed tablet orally, then intact tablet orally (Experimental): Single, 100 mg dose
  Interventions: Drug: BMS-986205
- BMS-986205 intact tablet orally then suspension via NG tube (Experimental): Single, 100 mg dose
  Interventions: Drug: BMS-986205
- BMS-986205 suspension via NG tube then intact tablet orally (Experimental): Single, 100 mg dose
  Interventions: Drug: BMS-986205

INTERVENTIONS:
Drug: BMS-986205 — Single 100 mg dose on Day 1 and Day 15

SUMMARY:
The purpose of this study is to evaluate the absorption of BMS-986205 into the bloodstream of healthy volunteers, when administered as an intact tablet taken orally, or as a crushed tablet taken orally with soft food, or as a crushed tablet suspension taken via a nasogastric (NG) tube. Eligible participants will be randomly assigned to 1 of 4 treatment sequences and will receive a single dose of BMS-986205 twice during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent form.
* Healthy male and female participants (not of childbearing potential), determined by no clinically significant deviation from normal in medical history, physical examination, ECGs (electrocardiograms) and clinical laboratory determinations.
* Women participants must have documented proof they are not of childbearing potential.
* Males sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for duration of treatment with BMS-986205, and for a total of 110 days after the last dose of BMS-986205; and must be willing to refrain from sperm donation during this time. Azoospermic males are exempt from contraceptive requirements.
* Normal renal function at screening (Glomerula Filtration Rate ≥ 80 mL/min/1.73 m2).
* Body Mass Index (BMI) of 18.0 kg/m2 to 32.0 kg/m2 inclusive.

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding.
* Any significant acute or chronic illness.
* Active tuberculosis (TB) requiring treatment, documented latent TB within the previous 3 years, or evidence of a past TB infection without documented adequate therapy. All participants will be required to have a QuantiFERON -TB Gold test performed at screening.
* History of Glucose-6-Phosphate Dehydrogenase deficiency (G6PD) or any other congenital hemolytic anemias.
* History of cardiac arrhythmias and/or autonomic instability.
* History of pulmonary, renal or liver disease.
* History of Gilbert's Syndrome.
* Recent (within 6 months of study drug administration) history of smoking or current smokers, including use of electronic cigarettes or nicotine-containing products such as tobacco for chewing, nicotine patches, nicotine lozenges or nicotine gum.
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo or psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger may enroll.
* Major surgery within 4 weeks of study drug administration.

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of single 100 mg dose of BMS-986205 administered orally as crushed tablet on soft food compared to intact tablet administered orally. | Up to 22 days
  Measured by plasma concentration.
Maximum observed plasma concentration (Cmax) of single 100 mg dose of BMS-986205 administered via nasogastric (NG) tube as crushed tablet suspension compared to intact tablet administered orally. | Up to 22 days
  Measured by plasma concentration.
Area under the plasma concentration time curve from time zero to 168 hours after dosing (AUC[0-168]) of single 100 mg dose of BMS-986205 administered orally as crushed tablet on soft food compared to intact tablet administered orally. | Up to 22 days
  Measured by plasma concentration.
Area under the plasma concentration time curve from time zero to 168 hours after dosing (AUC[0-168]) of single 100 mg dose of BMS-986205 administered via nasogastric (NG) tube as crushed tablet suspension compared to intact tablet administered orally. | Up to 22 days
  Measured by plasma concentration.

SECONDARY OUTCOMES:
Incidence of non-serious Adverse Events (AEs). | Up to 22 days
  Safety and tolerability as measured by incidence of non-serious AEs.
Incidence of Serious Adverse Events (SAEs). | Up to 22 days
  Safety and tolerability as measured by incidence of SAEs.
Number of participants with clinical laboratory abnormalities. | Up to 22 days
Number of participants with vital sign abnormalities. | Up to 22 days
Number of participants with electrocardiogram (ECG) abnormalities. | Up to 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Austin Clinic, Austin, Texas, United States

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx